CLINICAL TRIAL: NCT06915675
Title: The Adjunction of Flowable Decellularized Human Placental Connective Tissue Matrix in Alveolar Ridge Preservation: A Split Mouth Pilot Study
Brief Title: Human Placenta Extract Use in Socket Preservation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saint-Joseph University (Other)
Collaborators: Botiss Biomaterials GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: USJ-2024-175
Record Dates: First submitted 2025-03-28; First posted 2025-04-08 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Dental Extraction
Keywords: Alveolar ridge; Connective tissue; Extracellular matrix; Placental extracts; Wound healing; Tooth extraction
MeSH Terms: interventions — Placental Extracts; Transplantation, Homologous

STUDY DESIGN:
Intervention Model Description: Following the inclusion and exclusion criteria, 10 patients presenting a split mouth design will be enrolled in the study where one dental extraction site will serve as a test and the other will be the control
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placenta treatment arm (Active Comparator): Participants will receive allografts bone substitutes mixed with flowable human placental based connective tissue matrix in one extraction socket immediately following tooth extraction.
  Interventions: Biological: Placental Extract
- Control arm (Sham Comparator): Participants will receive allografts bone substitutes solely in one extraction socket immediately following tooth extraction.
  Interventions: Procedure: Allograft

INTERVENTIONS:
Biological: Placental Extract — Participants will receive allografts bone substitutes mixed with flowable human placental derived connective tissue matrix in one extraction socket immediately following tooth extraction.
  Arms: Placenta treatment arm
Procedure: Allograft — Participants will receive allografts bone substitutes solely in one extraction socket immediately following tooth extraction.
  Arms: Control arm

SUMMARY:
This split-mouth pilot study evaluates the effectiveness of flowable decellularized Human Placental Connective Tissue Matrix (HPCTM) in alveolar ridge preservation following tooth extraction. Patients will receive HPCTM mixed with allograft particles in one extraction socket and allograft particles solely in the contralateral socket. The primary outcome is to assess dimensional changes in the alveolar ridge in terms of soft tissue shrinkage using a super-imposed intra-oral scans taken at baseline , day 10, 21 and 30 post-op and bone resorption rate by comparing pre-op and 4 months post-op cone beam computed tomography scans. Secondary outcomes include clinical soft tissue healing evaluation and commentary. The HPCTM used in this study is regulated by the US FDA under Section 361 of the Public Health Service Act (21 CFR Part 1271.10(a)).

DETAILED DESCRIPTION:
- Data collection: The data collection process of the patients was divided into two steps: pre and post Alvealoar ridge preservation.

Before the surgery, clinical photographs using a digital single-lens reflex camera (Canon 90D, 100mm macro lens, Tokyo, Japan) equipped with a light diffuser (Flashkap, USA), CBCT and intra-oral scans of each patient were collected and stored separately.

After the surgery, the patients were asked to re-visit the dental clinic at 10,21 and 30 days post-operatively for a check-up, clinical photographs and intra-oral scans. Following a period of 4 months, the patients were again recalled to perform a CBCT scan and get sufficient information about the implant placement.

Surgical intervention:

All cases were performed by the same surgeon (B.H) who followed the same surgical protocol.

Following local anesthesia and crown removal if present (Fig. 1A,B) a minimally invasive cut using fissure carbide burrs (FG701, Neoburr, Republic of Korea) was performed to separate the mesial and distal roots. Subsequently the roots were luxated and extracted using elevators (EL3S, Hu-Friedy, USA) (Figure 1B, C). The alveolar sockets were debrided using Lucas curettes. Since avoiding blood inundation of the bone chips is not possible and to dodge any methodology biais, allografts were mixed with blood in both sites. The test sites received 0,5 cc of HCTM (Orafyl, Biocellgraft, USA) regulated by the US Food and Drug Administration (FDA) under Section 361 of the Public Health Service (HCT/P, 21 CFR, Part 1271.10(a) mixed with 0,5 cc of the patient's blood, the mixing procedure involved the use of a double syringes model with a mixing time of 2 minutes (Figure 2A). 1 cc of allografts particles (Maxgraft Cortico cancellous granules, Botiss, Germany) were mixed with the prepared serum continuously till a moldable putty was formed (Figure 2B). Subsequently, the bone putty was grafted in the socket and compacted softly till reaching the radiographic coronal limit of the socket (Figure 1F). Due to compaction process the excess of blood mixed with the gel filled the gingival portion of the socket resulting in a thick gelatinous seal of the socket. X shaped 5/0 Polytetrafluoroethylene sutures (Biotex, Purgo biologics, Republic of Korea) sutures were performed on the top of the socket to secure the grafted particles from spilling, care was giving to not displace the gingival margins of the socket (Figure 1H). The control socket received the same therapeutical treatment but with blood solely mixed to the allografts (Figure 1E) and a collagen fleece on top to prevent the bone particles from displacement (Figure 1G As a post-operative recommendation, the patients were advised to abstain from any gargling or spitting for 24 hours. The patients were given antibiotics for 7 days 2 g/day orally (Amoxicillin Sandoz®, Basel, Switzerland). Non-steroidal ani inflammatory drug ibuprofen 400 mg (Abbott Laboratories, Chicago, USA) three times daily for 3 days, and a chlorhexidine mouthwash (0.12%), three times daily for 2 weeks.

4 months post-op, a CBCT scan was performed to assess the bone dimensions and patients were recalled for implants placement. A full thickness flap was raised (Figure 3A) and implants (Blue diamond, Mega'gen, Republic of Korea) were placed in a prosthetically driven fashion making sure that the fixture was surrounded by at least 2 mm of bone buccally and lingually. Anatomical healing caps were used in order to sculpt an ideal prosthetic emergence profile (Figure 3B). Finally, two months later, a digital impression of the placed implant was performed using an intra-oral scan (R2I3, Mega'gen, Republic of Korea) and screw retained Zirconia crowns were delivered for each patient (Figure 3C, D).

-Studied parameters identification:

The studied parameters in this study were as follow:

1. Volumetric bone resorption rate expressed in %
2. Linear soft tissue shrinkage expressed in millimeters.
3. Clinical observation and interpretation of wound healing in test and control groups

2.5 Soft tissue healing measurements:

For an accurate and clear measurements several steps were followed; First all intra-oral scans were exported as a stereolithography file (STL). The initial intra-oral scans were imported to an imaging software and aligned to the CBCT scan using multiple stable landmarks, this scan was set as a reference, then they were exported to a design software (Medit Design, Medit, Republic of Korea) where teeth in relation were extracted virtually and the sockets filled till the top of the free gingiva. The follow-up intra-oral scans were imported to the same software and super-imposed using a semi-automatic option with up to 5 points were used as a stable reference. The region of interest was delimited using the trimming option as follow:

* Mesio-distally: 1,5 mm away from the concerned papilla peak.
* Apically: A bucco-lingual/palatal line tangent to the visible muco-gingival line and parallel to the occlusal surface.

Using the deviation analysis option of the software, a color map quantifying any positive or negative deviations between the different time points scans in comparison to the baseline was generated (Fig. 4).

2.6 Bone resorption measurements:

The hard tissue resorption measurement technique in a previous article published by the same authors was adopted 17. A semi-automatic segmentation software (ITK-Snap 4.0, U.S. National Institute of Biomedical Imaging and BioEngineering, USA) was used to load and segment the pre and post CBCT scans. First, both CBCTs were oriented according to the Frankfort plane, then aligned using multiple fixe landmarks in different orientations to ensure a perfect match and an easy reproducibility. A standard region of interest was applied for all the measured sites as follow:

A standard region of interest was applied for all the measured sites as follow:

* Mesio-distal limit: 1.5 mm away from the mesial and distal surface of adjacent tooth.
* Bucco-lingual limit: limited to the observed bone dimensions.
* Apico-coronal limit: Coronally the most detectable bone peak at the mesial and distal sides; apically, 1.5 mm below the root tip.

Using pixel-based scale, a specific threshold value was used to select and separate the desired structure from its surroundings of both pre and post-surgery CBCT. Following the automatic segmentations, a manual inspection was applied to eliminate any undesired selections and the volume of each created shape was measured using the software built-in tools (Fig. 5).

The resorption rate was calculated following the mathematical equation:

[ ( VPre-op-Vpost-op) / VPre-op] X 100.

Statistical analysis:

A descriptive statistical analysis was performed to describe the patient's characteristics. The data was expressed as the mean ± standard deviation. The Wilcoxon signed-rank test, a non-parametric test was deemed suitable for paired data and used to compare the volumetric bone resorption rate between the test (HPCTM + allograft) and control (allograft only) groups. As for the soft tissue shrinkage, paired t-test was applied to explore any statistical significance at day 10,21 and 30. Statistical significance was set at p < 0.05. All analyses were conducted using IBM SPSS Statistics 25.

ELIGIBILITY:
Inclusion Criteria:

* Age ranging between 20 and 60.
* Subjects having two hopeless teeth that needs extraction.
* Teeth fitting in the same morphological category (mono,bi or multirooted).
* Teeth belonging to different arch quadrants.
* Presence of more than half of the socket bone housing.
* Non-smoking patient.

Exclusion Criteria:

* Presence of active periodontal diseases i.e Miller class II and above categories.
* Presence of heavy metallic artefacts that can distort CBCT scans.
* Bad oral hygiene and non-compliance.
* Systemic diseases interfering with bone metabolism.
* Pregnant or lactating women.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2024-08-23 (Actual); Primary Completion 2025-02-11 (Actual); Study Completion 2025-04-10 (Estimated)

PRIMARY OUTCOMES:
Soft tisse shrinakge at different time points of the test and control groups | 30 days
  Using a measurement software ( Medit design, Medit, Republic of Korea) the intra-oral scans (.STL files) obtained at different time points of the healing process will be super-imposed and aligned. the following region of interest will be selected:
  * Mesio-distally: 1,5 mm away from the concerned papilla peak.
  * Apically: A bucco-lingual/palatal line tangent to the visible muco-gingival line and parallel to the occlusal surface.
  The deviation between the different scans which corresponds the soft tissue shrinkage will be automatically calculated in millimeters as a mean value with standard deviation
Bone resorption rate in test and control groups | 4 months
  . A semi-automatic segmentation software (ITK-Snap 4.0, U.S. National Institute of Biomedical Imaging and BioEngineering, USA) was used to load and segment the pre and post CBCT scans. First, both CBCTs were oriented according to the Frankfort plane, then aligned using multiple fixe landmarks in different orientations to ensure a perfect match and an easy reproducibility. A standard region of interest was applied for all the measured sites as follow:
  A standard region of interest was applied for all the measured sites as follow:
  * Mesio-distal limit: 1.5 mm away from the mesial and distal surface of adjacent tooth.
  * Bucco-lingual limit: limited to the observed bone dimensions.
  * Apico-coronal limit: Coronally the most detectable bone peak at the mesial and distal sides; apically, 1.5 mm below the root tip.
  Using pixel-based scale, a specific threshold value was used to select and separate the desired structure from its surroundings of both pre and post-surgery CBCT. Following the aut

SECONDARY OUTCOMES:
Clinical observation of the wound healing at control and test groups at 10, 21 and 30 days post-op | 30 days
  Before the surgery, clinical photographs using a digital single-lens reflex camera (Canon 90D, 100mm macro lens, Tokyo, Japan) equipped with a light diffuser (Flashkap, USA) of each patient were collected and stored separately.
  After the surgery, the patients were asked to re-visit the dental clinic at 10,21 and 30 days post-operatively for a check-up, clinical photographs and intra-oral scans.
  Same angulation photographs were stacked and an independent oral surgeon described the observed change in the alveolar tissues.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Joseph Younes, DDS,MSc, Phd, Study Director — Saint Joseph University of Beirut
Locations (1):
- Saint Joseph University of Beirut, Beirut, Beyrouth, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gulameabasse S, Gindraux F, Catros S, Fricain JC, Fenelon M. Chorion and amnion/chorion membranes in oral and periodontal surgery: A systematic review. J Biomed Mater Res B Appl Biomater. 2021 Aug;109(8):1216-1229. doi: 10.1002/jbm.b.34783. Epub 2020 Dec 22. PMID 33354857
- [Background] Kalsi AS, Kalsi JS, Bassi S. Alveolar ridge preservation: why, when and how. Br Dent J. 2019 Aug;227(4):264-274. doi: 10.1038/s41415-019-0647-2. PMID 31444438
- [Background] Chappuis V, Araujo MG, Buser D. Clinical relevance of dimensional bone and soft tissue alterations post-extraction in esthetic sites. Periodontol 2000. 2017 Feb;73(1):73-83. doi: 10.1111/prd.12167. PMID 28000281
- [Background] Chappuis V, Engel O, Reyes M, Shahim K, Nolte LP, Buser D. Ridge alterations post-extraction in the esthetic zone: a 3D analysis with CBCT. J Dent Res. 2013 Dec;92(12 Suppl):195S-201S. doi: 10.1177/0022034513506713. Epub 2013 Oct 24. PMID 24158340
- See also: Related Info — https://biocellgraft.com